CLINICAL TRIAL: NCT03532750
Title: Safety and Efficacy of Splenic Artery Embolization to Treat Symptomatic Portal
Brief Title: Splenic Embolization for Portal Hypertension
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD-2016-25151
Record Dates: First submitted 2018-04-25; First posted 2018-05-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Intervention Model Description: 1:1:1 randomization of participants in sequential order to either the control group (best medical management), particle embolization, and coil embolization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Control (No Intervention): This arm will undergo no study procedures and continue with best medical management. This entails managing pain and draining excess fluid.
- Particle (Experimental): Randomized to receive either the Embozene or Embosphere particles
  Interventions: Device: Particle
- Coil (Experimental): Randomized to receive either Ruby or Interlock detachable coils
  Interventions: Device: Coil

INTERVENTIONS:
Device: Particle — 1. 300-500 µm Embosphere Particles, Merit Medical (Rockland, MA) 501(k) number K991549.
  2. 300-500 µm Embozene Particles, Boston Scientific (Marlborough, MA) 501(k) number K133447.
  3. Ruby detachable coils, Penumbra (Alameda, CA) 501(K) number K103305.
  4. Interlock detachable coils, Boston Scientific (Marlborough, MA) 501(k) number K132578.
  Other Names: Embosphere Particles; Embozene Particles
  Arms: Particle
Device: Coil — Ruby or Interlock detachable coils
  Other Names: Ruby Detachable Coils; Interlock Detachable Coils
  Arms: Coil

SUMMARY:
The primary purpose of this study is to evaluate the safety and efficacy of partial splenic artery embolization in the treatment of symptomatic portal vein hypertension. A secondary aim is to evaluate the relative efficacy of two separate splenic artery embolization techniques, coiling versus particle embolization of the spleen. These two methods will be compared to standard medical management which consist of pain management and fluid draining.

DETAILED DESCRIPTION:
This is a single center phase I/II study that is designed to assess the safety and efficacy of splenic artery embolization in the setting of symptomatic portal hypertension. All participating investigators have signed the protocol agreement and no investigator will be added until they sign the agreement. The study will not be initiated until FDA and IRB approval is obtained.

The study will consist of a 4 week screening period, day of treatment, and 12-month follow-up period. 60 subjects will be enrolled, with a goal of randomizing 30, at the University of Minnesota Medical Center. Enrollment is expected to take up to 48 months. The collection of data will be accomplished by utilizing a clinical research team that will obtain symptomatic portal hypertension improvement and safety assessments. Efficacy assessments will include; change in portal vein velocity, ascitic fluid production change, reduction in splenic size, and improvement in quality of life (QoL). Safety assessments include subject and investigator reported adverse events, subjective pain, and splenic abscess formation.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are between 22-70 years of age.

  * Patient must have portal hypertension; as defined by: refractory ascites or unilateral right sided pleural effusions with concomitant liver cirrhosis and splenomegaly (spleen > 11 cm on CT or US).
  * Medically refractive/intolerant, ascites or unilateral right sided pleural effusions consistent with hepatic hydrothorax. Medically refractive defined as those with persistent need for paracentesis or thoracentesis despite maximal doses of diuretics (400 mg spironolactone and 160 mg furosemide per day) or those who are intolerant of furosemide (develop azotemia, electrolyte imbalance, encephalopathy or renal failure) or spironolactone (develop gynecomastia, decreased libido, and hyperkalemia).
  * Patients will need to meet one or more of the following requirements:

    * MELD >18 but <35
    * Anatomic variation making TIPS impossible/difficult
    * Previous failed attempt to place TIPS
    * Unwilling to undergo TIPS
    * History of severe hepatic encephalopathy
    * Thrombosis of the hepatic veins
  * Willing and able to provide informed consent

Exclusion Criteria:

* Patients < 22 and >70 years of age
* Patients with CLDQ score of >6 or <2
* Patients with a weight >400 pounds
* Patients with primary or secondary splenic cancer
* Currently pregnant
* Current systemic infection
* Patients who have undergone prior splenectomy or other splenic surgery
* Patients who have previously undergone splenic artery embolization for any reason (likely reasons would be trauma or thrombocytopenia)
* Patients with splenic vascular anatomy that would increase the risk of non-target embolization.
* Patients who have a INR or platelet count which are not correctable to <1.8 and >35,000 respectively
* Anaphylaxis to intravenous contrast.
* Patients diagnosed with Budd-Chiari Syndrome (This will be assessed on pre-intervention CTA)

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | pre-procedural (baseline) and at 1, 3, 6, and 12 month follow-up visits
  Administration of the Chronic Liver Disease Questionnaire (CLDQ)
Incidence of Treatment Adverse Events | Patients will be evaluated for adverse events post procedural at 72hrs, 1 week, and 1, 3, 6, and 12 months
  Evaluation of all procedure-related adverse events (PRAE) and serious adverse events (SAE)

SECONDARY OUTCOMES:
Ascites Production | pre-procedural and at 1, 3, and 6 months
  Fluid production
Splenic Size | pre-procedural and at 1,3,6 and 12 months
  Changes in size of spleen as indicated by MRI or CT
Portal Vein Velocity | pre-procedural and at 1, 6 and 12 months
  Changes in flow volume and velocity as evidenced by ultra sound

CONTACTS AND LOCATIONS:
Overall Officials: Shamar Young, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
All IPD generated for this study will only be reviewed by the study personnel who have been approved by the IRB. Any results that are shared, will be aggregate group data that does not address any individual participant directly.